CLINICAL TRIAL: NCT01525810
Title: A Long-Term Follow-Up Study of Subjects Who Participated in a Clinical Trial in Which Peginterferon Lambda-1a (BMS-914143) Was Administered for the Treatment of Chronic Hepatitis C
Brief Title: Three-year Follow-up Study of Subjects Who Participated in a Previous Lambda (BMS-914143) Chronic Hepatitis C Clinical Trial
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI452-016; 2011-005293-31 (EudraCT Number)
Record Dates: First submitted 2012-01-11; First posted 2012-02-03 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects treated with Peginterferon Lambda-1a (BMS-914143): Subjects who participated in a clinical trial in which Peginterferon Lambda-1a (BMS-914143) was administered for the treatment of chronic hepatitis C
  Interventions: Drug: Peginterferon Lambda-1a (BMS-914143)

INTERVENTIONS:
Drug: Peginterferon Lambda-1a (BMS-914143) — Observational study - No Intervention [subjects were previously treated with Peginterferon Lambda-1a (BMS-914143)]

SUMMARY:
The primary purpose of this study is to determine whether the hepatitis C virus continues to remain unable to be detected in subjects who were previously treated with BMS-914143 and achieved sustained virologic response

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have received Lambda in a previous trial and have Hepatitis C virus (HCV) Ribonucleic acid (RNA) < LOQ at the completion of the required post-treatment follow-up (must enter this study within 6 months of completion of the required post-treatment follow-up in the previous trial) NOTE: For blinded parent trials, subjects who have HCV RNA <LOQ at the completion of the required post-treatment follow-up may enter this study without knowledge of their treatment assignment in the parent study. Subjects who received control agents (eg, pegylated-interferon alfa) in the previous protocol will be allowed to participate until unblinded treatment information is released; at that time subjects will have the option to continue in the study

Exclusion Criteria:

* Subjects must not have been treated with any antiviral or immunomodulatory drug for chronic hepatitis C after completion of the previous study of Lambda

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who participated in a clinical trial in which BMS-914143 was administered for the treatment of chronic hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Durability of virologic response (time to loss of virologic response) | 24 week intervals from end of treatment in parent study up to 144 weeks
  Durability of virologic response as assessed by the time to loss of virologic response in subjects treated in a previous study with BMS-914143 who have HCV RNA less than the limit of quantitation of the assay (< LOQ) at the completion of the required post-treatment follow-up in the previous study. Loss of virologic response assessed using HCV RNA at 24-week intervals

SECONDARY OUTCOMES:
Long-term progression of liver disease | 24 week intervals up to 144 weeks
  Long-term progression of liver disease as measured by laboratory indicators of hepatic status and function, all-cause mortality and liver related mortality in subjects previously treated with BMS-914143 who have HCV RNA < LOQ at the completion of the required post-treatment follow-up in the parent study
Duration of persistence of anti-Lambda antibodies in subjects who are positive for anti-Lambda antibodies at end of treatment in the parent study | 24 week intervals up to 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (69):
- United States (17):
  - Scripps Clinic, La Jolla, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Orlando Immunology Center, Orlando, Florida
  - Gastrointestinal Specialists Of Georgia, Marietta, Georgia
  - The Queen'S Medical Center, Honolulu, Hawaii
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Consultants For Clinical Research, Cincinnati, Ohio
  - Texas Clinical Research Institute, Arlington, Texas
  - St. Luke'S Episcopal Hospital - Baylor College Of Medicine, Houston, Texas
  - University Of Texas Health Science Center At Houston, Houston, Texas
  - Va Medical Center (151), Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Clinical Research Centers Of America, Murray, Utah
  - Metropolitan Research, Annandale, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Buenos Aires
- Australia (13):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution, Sydney, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Herston, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Parkville, Victoria
- Local Institution, Vienna, Austria
- Belgium (2):
  - Local Institution, Leuven
  - Local Institution, Liège
- Toronto Digestive Disease Associates, Inc., Vaughan, Ontario, Canada
- Local Institution, Hus, Finland
- France (6):
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pessac
- Germany (2):
  - Local Institution, Hamburg
  - Local Institution, Heidelberg
- Greece (2):
  - Local Institution, Athens
  - Local Institution, Thessaloniki
- Italy (6):
  - Local Institution, Cisanello (pisa)
  - Local Institution, Florence
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Novara
  - Local Institution, Viale Del Policlinico, 155
- Local Institution, Guadalajara, Jalisco, Mexico
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Leiden
- Local Institution, Auckland, New Zealand
- Poland (3):
  - Local Institution, Bialystok
  - Local Institution, Krakow
  - Local Institution, Wroclaw
- Local Institution, San Juan, Puerto Rico
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Iași
  - Local Institution, Timișoara
- Local Institution, Busan, South Korea
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Valencia

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx